CLINICAL TRIAL: NCT03371771
Title: Volunteer-Delivery of Behavioral Activation for Senior Center Clients
Brief Title: Volunteer-Delivery of Behavioral Activation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Patrick Raue, Professor, School of Medicine: Psychiatry: Population Health, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00002543; R34MH111849 (NIH)
Record Dates: First submitted 2017-12-08; First posted 2017-12-13 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive either Volunteer or MSW-delivered Behavioral Activation
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Volunteer-delivered Behavioral Activation (Experimental)
  Interventions: Behavioral: Volunteer-delivered Behavioral Activation
- MSW-delivered Behavioral Activation (Active Comparator)
  Interventions: Behavioral: MSW-delivered Behavioral Activation

INTERVENTIONS:
Behavioral: Volunteer-delivered Behavioral Activation — Behavioral Activation as delivered by trained volunteers
  Arms: Volunteer-delivered Behavioral Activation
Behavioral: MSW-delivered Behavioral Activation — Behavioral Activation as delivered by trained MSWs
  Arms: MSW-delivered Behavioral Activation

SUMMARY:
In response to large numbers of senior center clients who suffer untreated depression and the dearth of geriatric mental health providers, the investigators have simplified a Behavioral Activation intervention to match the skill set of age-matched lay volunteers available to senior centers (Volunteer BA). This R34 proposes developmental work on delivering Volunteer BA in senior centers, so as to arrive to a sustainable intervention with standardized procedures. The investigators follow with a small randomized controlled trial (RCT) testing the comparative impact of Volunteer BA versus MSW-provided BA on increased client activity and reduced depressive symptoms.

DETAILED DESCRIPTION:
Senior centers provide social, health, nutritional, and recreational services to older adults. Ten percent of older adults in these settings experience clinically significant depression. Although many aging services now screen for depressive symptoms, an IOM report indicates that the number of geriatric mental health providers nationally is insufficient. Further complicating treatment delivery is the reluctance of depressed elders to accept a mental health referral or pursue treatment. It has been proposed that lay workers may be able to offer psychosocial interventions for geriatric mental health disorders. Lay volunteer-delivered interventions may improve depression outcomes, may do so by engaging the same target variables as professionally-delivered interventions, and may be both more cost effective and acceptable to seniors. Limitations include uncertainties about training and supervision needs, reliable methods to assure intervention fidelity and patient safety, and comparability of outcomes to those attained by professionally- delivered interventions. Building on senior centers' volunteer programs, this proposal utilizes senior volunteers to meet the mental health needs of depressed urban clients. To this end, the investigators simplified Behavioral Activation (BA) to match the skill set of lay senior volunteers (Volunteer BA). The investigators chose BA because it is an effective treatment for late-life depression, can be administered by paraprofessionals, and its primary mechanism (target) of action has been validated by efficacy studies. Based on preliminary data, the investigators aim to test the feasibility and acceptability of Volunteer BA for an underserved and difficult to engage population. The investigators propose further developmental work on the delivery of Volunteer BA in senior centers, so as to arrive at a sustainable intervention with standardized procedures. The investigators propose a small RCT testing the impact of Volunteer BA versus MSW-delivered standard BA on increased client activity (the target) and reduced depressive symptoms (clinical outcome). The Volunteer BA delivery model: 1. Makes use of existing volunteer resources; 2. has potential for being an acceptable and sustainable intervention; and 3. is expected to engage BA targets. However, its capacity to yield comparable outcomes to MSW-delivered BA is yet to be determined.

ELIGIBILITY:
Inclusion Criteria:

Referral to study (stage 1):

1. Age ≥ 60 years.
2. Attends one of 4 participating Seattle senior centers.
3. PHQ-9 score of ≥10 via routine screening.

Research assessment (stage 2):

1. Mini Mental State Exam (MMSE) ≥ 24.
2. Capacity to provide written consent for both research assessment and the BA intervention.

Exclusion Criteria:

1. Current passive or active suicidal ideation (SCID-V or HAM-D).
2. Presence of psychiatric diagnoses other than unipolar, non-psychotic major depression or anxiety disorder by SCID-V.
3. Severe or life-threatening medical illness (e.g., end stage organ failure).
4. Inability to speak English.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Behavioral Activation for Depression Scale (BADS) scores | Baseline and 9 weeks
  The Behavioral Activation for Depression Scale (range 0-150; higher scores indicate higher levels of activation) change score from baseline to 9 weeks
Change from Baseline in Hamilton Rating Scale for Depression (HAM-D) scores | Baseline and 9 weeks
  Hamilton Depression Rating Scale for Depression (range 0-76; higher scores indicate greater severity of depression) change score from baseline to 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Patrick J Raue, PhD, Principal Investigator — University of Washington
Locations (4):
- United States (4):
  - Greenwood Senior Center, Seattle, Washington
  - Wallingford Senior Center, Seattle, Washington
  - Southeast Senior Center, Seattle, Washington
  - Central Area Senior Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No